CLINICAL TRIAL: NCT02863965
Title: High Definition Endoscopy and Optic Enhancement Endoscopy in Gastric Neoplasia: A Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2016SDU-QILU-13
Record Dates: First submitted 2016-07-30; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Gastric Neoplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- High definition endoscopy and optic enhancement: All the patients underwent routine preparation before the procedure. The detected lesions in high definition endoscopy were observed with optic enhancement mode. The endoscopist was required to give the real-time descriptions of surface pit patterns of the lesions, based on surface pattern classification. After that, biopsy specimens will be obtained respectively by forceps from each detected lesion recorded for histologic diagnosis.

SUMMARY:
The aim of the study is to evaluate the diagnostic value of high definition endoscopy and optic enhancement in gastric neoplasia.

ELIGIBILITY:
Inclusion Criteria:

* patients with dyspeptic symptoms and aged 40 years or older
* or patients with Helicobacter pylori infection, or histologically verified gastric intestinal metaplasia or atrophic gastritis
* or patients with family history of gastric cancer

Exclusion Criteria:

* presence of gastrectomy, acute gastrointestinal bleeding, or known gastric neoplasia
* presence of conditions unsuitable for endoscopy procedure including coagulopathy, impaired cardiopulmonary function , pregnancy or breastfeeding
* inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dyspeptic symptoms and aged 40 years or older, or with Helicobacter pylori infection, histologically verified gastric intestinal metaplasia or atrophic gastritis, or with family history of gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of optical enhancement endoscopy in diagnosis of gastric neoplasia | 8 months
Specificity of optical enhancement endoscopy in diagnosis of gastric neoplasia | 8 months
Positive predictive value of optical enhancement endoscopy in diagnosis of gastric neoplasia | 8 months
Negative predictive value of optical enhancement endoscopy in diagnosis of gastric neoplasia | 8 months

SECONDARY OUTCOMES:
The inter-observer and intra-observer agreement of optic enhancement endoscopy in gastric neoplasia | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD. MD., Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China